CLINICAL TRIAL: NCT02586883
Title: Study of the Bronchial Trans-epithelial Transport in Patients With Idiopathic Multiple Dilations of the Bronchi
Brief Title: Bronchial Trans-epithelial Transport in Patients With Idiopathic Multiple Dilations of the Bronchi
Acronym: EPITRANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00731-48
Record Dates: First submitted 2015-07-13; First posted 2015-10-27 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Idiopathic Dilation of the Bronchi
Keywords: Dilation of the Bronchi; Bronchial potential difference; Dilation of the Bronchi (DDB)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with multiple bronchi dilations (Experimental)
  Interventions: Other: bronchial ddp test
- Control patients without transport abnormality (Active Comparator)
  Interventions: Other: bronchial ddp test
- Patients with typical cystic fibrosis (Active Comparator)
  Interventions: Other: bronchial ddp test

INTERVENTIONS:
Other: bronchial ddp test — bronchial ddp test during endoscopy, nasal smear, bronchial smear

SUMMARY:
The purpose of this study is to identify the abnormalities of bronchial trans-epithelial transport of chloride, sodium and bicarbonate in patients with idiopathic dilations of the bronchi.

DETAILED DESCRIPTION:
Dilations of the bronchi happens for one child over 3000. The extended forms may progress to respiratory failure. More than one case over two remains of undetermined cause. If the prototype is the cystic fibrosis, other abnormalities of ionic transport may be the cause of a failure of mucociliary clearance and enhance the idiopathic dilations of the bronchi.

The purpose of this study is to identify the abnormalities of bronchial trans-epithelial transport of chloride, sodium and bicarbonate in patients with idiopathic dilations of the bronchi, in comparison to two others groups of patients (without abnormality of ionic transport/with typical cystic fibrosis).

ELIGIBILITY:
Inclusion Criteria:

Common criteria for all patients

* Age between 2 and 20 years.
* Patient weighing more than 12kg
* Patients with a scheduled bronchoscopy under clinical monitoring (assessment of bronchial involvement, local samples for bacteriological and histological examination)
* Signature of consent by the patient or by the / the holder (s) of parental authority and the investigator
* Patient affiliated to a social security scheme or entitled
* Patient with contraception (for woman of childbearing age) Specific criteria for idiopathic bronchiectasis patients Patient with idiopathic bronchiectasis in at least two lobes, diagnosis made after extensive screening of known acquired or congenital causes

Specific criteria for "control" patients without abnormal ion transport

* Patient Not having bronchiectasis s or any supposed alteration in transepithelial ion transport
* Patients with fiberoptic bronchoscopy performed for one of the following indications:
* Pulmonary malformations
* Laryngeal, tracheal, bronchomalacia
* Airway compression
* Interstitial pathology
* Suspicion of foreign body
* Suspected tuberculosis Specific criteria for patients with a typical form of cystic f ibrosis (CF) Patient carrying 2 causing mutations in the CFTR gene (according to CFTR2 database; http://www.cftr2.org/mutations_history.php) and sweat test> 60 milliequivalent per liter (mEq/L).

Exclusion Criteria:

Common criteria for all patients

* Smoking passive or active
* Not essential bronchial endoscopy in the clinical follow
* Extension of bronchoscopy time attributed to the difference in potential bronchial incompatible with the patient's general status
* Patient pregnant or breast feeding
* Hypersensitivity or cons known contraindications to health products for measurement of DDP (isoproterenol, Amiloride, ATP)

Specific criteria for idiopathic DDB patients

Presence of other congenital or acquired etiologies of DDB:

* Typical or atypical cystic fibrosis,
* Immunodeficiency,
* Primary ciliary dyskinesia,
* Abnormal bronchial wall structure (Williams-Campbell syndrome, Mounier-Kuhn, Ehlers-Danlos syndrome, Marfan's disease)
* Infectious DDBs post
* Extrinsic or endobronchial obstruction (foreign body, malformation, middle lobe syndrome)
* Chronic inhalation (GERD, swallowing disorders, gastroesophageal tracheal fistula)
* Allergic bronchopulmonary aspergillosis,
* System disease.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Response to isoproterenol in solution without chloride ions during bronchial potential difference test (ΔIsoprotérénol / bronchial). | up to 5 days
  Difference between groups for Level of repolarisation

SECONDARY OUTCOMES:
Response to amiloride during bronchial potential difference test | up to 5 days
  Trans-epithelial transport measured in vivo
trans-epithelial ionic transport in the nasal epithelium (nasal DDP) | up to 5 days
  Trans-epithelial transport measured in vivo
trans-epithelial ionic transport of sweat epithelium (sweat test) | up to 5 days
  Trans-epithelial transport measured in vivo
Basal current short circuit | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Response to Epithelial Sodium Channel (ENaC) inhibitors | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Activation of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Inhibition of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) (inh-172) | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Activation of Calcium (Ca)-dependent Chloride (Cl-) ion channels | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Inhibition of Solute Carrier family 26, member 9 (SLC26A9) | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Response to inhibitors of potassium (K+ ) secretion basolateral | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures
Bicarbonate (HCO3- ) secretion in response to forskolin | up to 5 days
  Trans-bronchial epithelial ionic transport evaluated in vitro on bronchial primary cultures

CONTACTS AND LOCATIONS:
Locations (1):
- Necker-Enfants Malades Hospital, Paris, France